CLINICAL TRIAL: NCT02690181
Title: A Phase 2, Non-Randomized, Controlled, Open-Label, Parallel-Group, Extension Study to Evaluate the Immunogenicity and Safety of the Second Dose of GBS Trivalent Vaccine in Healthy Non-pregnant Subjects.
Brief Title: Extension Study to Evaluate the Immunogenicity and Safety of the Second Dose of GBS Trivalent Vaccine in Healthy Non-Pregnant Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205421; 2015-003094-15 (EudraCT Number); V98_06E1 (Other: Novartis)
Record Dates: First submitted 2016-02-16; First posted 2016-02-24 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Bacterial Infection Due to Streptococcus, Group B; Streptococcus Agalactiae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- GBS NoAdj/GBS NoAdj (Experimental): Subjects who had received unadjuvanted GBS Trivalent Vaccine in parent study V98_06 (205468 - NCT01150123) and received a single dose of unadjuvanted GBS Trivalent Vaccine in V98_06E1 (205421 - NCT02690181).
  Interventions: Biological: GBS Trivalent Vaccine
- GBS Alum/GBS NoAdj (Experimental): Subjects who had received GBS Trivalent Vaccine with alum adjuvant in parent study V98_06 (205468 - NCT01150123) and received a single dose of unadjuvanted GBS Trivalent Vaccine in V98_06E1 (205421 - NCT02690181).
  Interventions: Biological: GBS Trivalent Vaccine
- GBS MF59 Full/GBS NoAdj (Experimental): Subjects who had received GBS Trivalent Vaccine with full dose of MF59 in parent study V98_06 (205468 - NCT01150123) and received a single dose of unadjuvanted GBS Trivalent Vaccine in V98_06E1 (205421 - NCT02690181).
  Interventions: Biological: GBS Trivalent Vaccine
- GBS MF59 Half/GBS NoAdj (Experimental): Subjects who had received GBS Trivalent Vaccine with half dose of MF59 in parent study V98_06 (205468 - NCT01150123) and received a single dose of unadjuvanted GBS Trivalent Vaccine in V98_06E1 (205421 - NCT02690181).
  Interventions: Biological: GBS Trivalent Vaccine
- Placebo/GBS NoAdj (Experimental): Subjects who had received placebo in parent study V98_06 (205468 - NCT01150123) and received a single dose of unadjuvanted GBS Trivalent Vaccine in V98_06E1 (205421 - NCT02690181).
  Interventions: Biological: GBS Trivalent Vaccine
- Naive/GBS NoAdj (Experimental): Healthy non-pregnant female subjects aged 22 through 46 years inclusive on the day of informed consent who had not received any GBS vaccine in the past and who received a single dose of unadjuvanted GBS Trivalent Vaccine in V98_06E1 (205421 - NCT02690181).
  Interventions: Biological: GBS Trivalent Vaccine

INTERVENTIONS:
Biological: GBS Trivalent Vaccine — Administration of lyophilized formulation of a GBS trivalent vaccine containing 5 µg of each polysaccharide capsules from serotypes Ia, Ib, and III of Group B Streptococcus conjugated to CRM-197 .

SUMMARY:
The objective of this extension study is the initial assessment of safety and immunogenicity of the second dose of GBS Trivalent Vaccine following the time interval that is close to the inter-pregnancy interval observed in the general population.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-pregnant subjects who have received a single 5 µg dose of GBS Trivalent Vaccine or placebo in the V98_06 study and healthy non-pregnant female subjects aged 22-46 years inclusive on the day of informed consent who have not received any GBS vaccine in the past
2. Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator
3. Females of childbearing potential who are using an effective birth control method which they intend to use until the end of the study (day 181 visit) or females of non-childbearing potential

Exclusion Criteria:

1. Progressive, unstable or uncontrolled clinical conditions, or clinical conditions representing a contraindication to intramuscular vaccination and blood draws
2. Abnormal function of the immune system
3. Received immunoglobulins or any blood products within 180 days prior to informed consent
4. Received an investigational or non-registered medicinal product within 30 days prior to informed consent
5. Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study
6. Individuals who received any other vaccines within 14 days for inactivated vaccines or 28 days for live vaccines prior to enrolment in this study or who are planning to receive any vaccine within 28 days from the study vaccination. Exception - an inactivated influenza vaccine may be administered up to 7 days prior to study vaccination or 7 days after study vaccination
7. Individuals who anticipate becoming pregnant prior to the end of the study, or individuals who are breastfeeding
8. Individuals who have had a previous immunization with a vaccine containing Group B Streptococcus antigens that was not part of V98_06 study
9. Individuals with a fever (oral temperature ≥ 38°C) within 3 days prior to day 1 or use of antipyretics and/or analgesic medications within 24 hours prior to day 1
10. Individuals with acute or chronic infection(s) that require systemic antibiotic treatment or antiviral therapy, within 7 days prior to day 1

Ages: 22 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2016-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20047

REFERENCES:
- [Background] Leroux-Roels G, Bebia Z, Maes C, Aerssens A, De Boever F, Grassano L, Buffi G, Margarit I, Karsten A, Cho S, Slobod K, Corsaro B, Henry O. Safety and Immunogenicity of a Second Dose of an Investigational Maternal Trivalent Group B Streptococcus Vaccine in Nonpregnant Women 4-6 Years After a First Dose: Results From a Phase 2 Trial. Clin Infect Dis. 2020 Jun 10;70(12):2570-2579. doi: 10.1093/cid/ciz737. PMID 31394574

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 site in Belgium.
Pre-assignment Details: All enrolled subjects completed the study.
Groups:
- GBS NoAdj/GBS NoAdj Group: Subjects who had received unadjuvanted GBS Trivalent Vaccine in parent study V98_06 (205468 - NCT01150123) and received a single dose of unadjuvanted GBS Trivalent Vaccine in V98_06E1 (205421 - NCT02690181).
- GBS Alum/GBS NoAdj Group: Subjects who had received GBS Trivalent Vaccine with alum adjuvant in parent study V98_06 (205468 - NCT01150123) and received a single dose of unadjuvanted GBS Trivalent Vaccine in V98_06E1 (205421 - NCT02690181).
- GBS MF59 Half/GBS NoAdj Group: Subjects who had received GBS Trivalent Vaccine with half dose of MF59 in parent study V98_06 (205468 - NCT01150123) and received a single dose of unadjuvanted GBS Trivalent Vaccine in V98_06E1 (205421 - NCT02690181).
- GBS MF59 Full/GBS NoAdj Group: Subjects who had received GBS Trivalent Vaccine with full dose of MF59 in parent study V98_06 (205468 - NCT01150123) and received a single dose of unadjuvanted GBS Trivalent Vaccine in V98_06E1 (205421 - NCT02690181).
- Placebo/GBS NoAdj Group: Subjects who had received placebo in parent study V98_06 (205468 - NCT01150123) and received a single dose of unadjuvanted GBS Trivalent Vaccine in V98_06E1 (205421 - NCT02690181).
- Naive/GBS NoAdj Group: Healthy non-pregnant female subjects aged 22 through 46 years inclusive on the day of informed consent who had not received any GBS vaccine in the past and who received a single dose of unadjuvanted GBS Trivalent Vaccine in V98_06E1 (205421 - NCT02690181).
Period: Overall Study
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Started | 14 | 14 | 15 | 10 | 6 | 21
Completed | 14 | 14 | 15 | 10 | 6 | 21
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group | Total
Number analyzed (Participants) | 14 | 14 | 15 | 10 | 6 | 21 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.4 (6.91) | 31.6 (6.06) | 28.9 (4.68) | 29.7 (6.22) | 28.3 (5.39) | 29.2 (6.96) | 30.1 (6.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 15 | 10 | 6 | 21 | 80
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 14 | 15 | 10 | 6 | 21 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With ELISA Antibody Concentrations of GBS Serotype Ia Above Pre-specified Thresholds - Day 61
Description: Percentage of subjects who reach pre-defined sequential serotype-specific serum antibody levels for serotype Ia at Day 61 post-vaccination, as measured by Enzyme-linked immunosorbent Assay (ELISA).
Time Frame: At Day 61
Population: All screened subjects who provided informed consent and baseline screening measurements, received a subject ID, received study vaccine according to the protocol, and parent study vaccine (non-naïve subjects), and provided immunogenicity data at Day 1, Day 31 or Day 61 in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 13 | 14 | 15 | 10 | 5 | 20
Percentage of subjects
  ≥ 0.1 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [47.8 to 100] | 100 [83.2 to 100]
  ≥ 0.2 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [47.8 to 100] | 95 [75.1 to 99.87]
  ≥ 0.5 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [47.8 to 100] | 90 [68.3 to 98.8]
  ≥ 1 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 80 [28.4 to 99.5] | 85 [62.1 to 96.8]
  ≥ 2 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 60 [14.7 to 94.7] | 65 [40.8 to 84.6]
  ≥ 3 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 93 [68.1 to 99.83] | 90 [55.5 to 99.75] | 60 [14.7 to 94.7] | 60 [36.1 to 80.9]
  ≥ 5 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 93 [68.1 to 99.83] | 90 [55.5 to 99.75] | 60 [14.7 to 94.7] | 60 [36.1 to 80.9]
  ≥ 8 µg/mL | 92 [64 to 99.81] | 100 [76.8 to 100] | 93 [68.1 to 99.83] | 90 [55.5 to 99.75] | 60 [14.7 to 94.7] | 60 [36.1 to 80.9]

2. Primary Outcome: Percentage of Subjects With Antibody Concentrations of GBS Serotype Ib Above Pre-specified Thresholds - Day 61
Description: Percentage of subjects who reach pre-defined sequential serotype-specific serum antibody levels for serotype Ib at day 61 post-vaccination. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 61
Population: All screened subjects who provided informed consent and baseline screening measurements, received a subject ID, received study vaccine according to the protocol, and parent study vaccine (non-naïve subjects), and provided immunogenicity data at Day 1, Day 31 or Day 61 in this study.in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 13 | 14 | 15 | 10 | 5 | 20
Percentage of subjects
  ≥ 0.1 μg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [47.8 to 100] | 85 [62.1 to 96.8]
  ≥ 0.2 μg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [47.8 to 100] | 80 [56.3 to 94.3]
  ≥ 0.5 μg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 80 [28.4 to 99.5] | 70 [45.7 to 88.1]
  ≥ 1 μg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 60 [14.7 to 94.7] | 65 [40.8 to 84.6]
  ≥ 2 μg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 60 [14.7 to 94.7] | 50 [27.2 to 72.8]
  ≥ 3 μg/mL | 100 [75.3 to 100] | 93 [66.1 to 99.82] | 100 [78.2 to 100] | 100 [69.2 to 100] | 60 [14.7 to 94.7] | 50 [27.2 to 72.8]
  ≥ 5 μg/mL | 85 [54.6 to 98.1] | 93 [66.1 to 99.82] | 100 [78.2 to 100] | 100 [69.2 to 100] | 60 [14.7 to 94.7] | 45 [23.1 to 68.5]
  ≥ 8 μg/mL | 85 [54.6 to 98.1] | 93 [66.1 to 99.82] | 93 [68.1 to 99.83] | 100 [69.2 to 100] | 20 [0.5 to 71.6] | 40 [19.1 to 63.9]

3. Primary Outcome: Percentage of All Subjects With Antibody Concentrations of GBS Serotype III Above Pre-specified Thresholds - Day 61
Description: Percentage of subjects who reach pre-defined sequential serotype-specific serum antibody levels for serotype III at day 61 post-vaccination. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 61
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 13 | 13 | 15 | 10 | 5 | 20
Percentage of subjects
  ≥ 0.1 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [47.8 to 100] | 100 [83.2 to 100]
  ≥ 0.2 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [47.8 to 100] | 80 [56.3 to 94.3]
  ≥ 0.5 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 80 [28.4 to 99.5] | 80 [56.3 to 94.3]
  ≥ 1 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 40 [5.3 to 85.3] | 75 [50.9 to 91.3]
  ≥ 2 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 40 [5.3 to 85.3] | 65 [40.8 to 84.6]
  ≥ 3 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 40 [5.3 to 85.3] | 65 [40.8 to 84.6]
  ≥ 5 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 40 [5.3 to 85.3] | 50 [27.2 to 72.8]
  ≥ 8 μg/mL | 100 [75.3 to 100] | 92 [64 to 99.81] | 100 [78.2 to 100] | 100 [69.2 to 100] | 40 [5.3 to 85.3] | 50 [27.2 to 72.8]

4. Primary Outcome: Numbers of Subjects With Solicited Local and Systemic Adverse Events (AEs)
Description: Threshold for Erythema, Swelling and Induration: None (0 mm), Any (>= 1 mm).
Time Frame: Day 1 to Day 7
Population: All screened subjects who signed informed consent form, provided demographic data and/or baseline screening assessments, were randomized and assigned a study subject ID, received the study vaccination and with any solicited adverse event data and/or indicators of solicited adverse events (e.g., use of analgesics/antipyretics).
Measure: Count of Participants; unit: Participants
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 14 | 14 | 15 | 10 | 5 | 21
Participants
  Any Local | 11 | 12 | 10 | 6 | 3 | 11
  Pain | 10 | 9 | 9 | 6 | 3 | 11
  Erythema | 1 | 4 | 2 | 1 | 1 | 3
  Swelling: number analyzed (Participants) | 14 | 14 | 15 | 10 | 5 | 20
  Swelling | 0 | 2 | 4 | 1 | 1 | 0
  Warmth | 1 | 4 | 4 | 2 | 2 | 2
  Induration: number analyzed (Participants) | 14 | 14 | 15 | 10 | 5 | 20
  Induration | 2 | 2 | 5 | 2 | 1 | 0
  Ecchymosis: number analyzed (Participants) | 14 | 14 | 15 | 10 | 5 | 20
  Ecchymosis | 0 | 0 | 1 | 0 | 0 | 1
  Any Systemic | 5 | 11 | 7 | 5 | 2 | 5
  Chills | 0 | 0 | 1 | 1 | 1 | 0
  Nausea | 0 | 2 | 2 | 0 | 0 | 1
  Malaise | 0 | 2 | 2 | 2 | 1 | 1
  Generalized Myalgia | 2 | 2 | 2 | 1 | 1 | 1
  Generalized Arthralgia | 0 | 1 | 2 | 0 | 0 | 0
  Headache | 4 | 4 | 5 | 2 | 2 | 4
  Fatigue | 3 | 10 | 4 | 4 | 1 | 2
  Body Rash | 0 | 1 | 0 | 0 | 0 | 0
  Fever (≥ 38°C) | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: The number of subjects with any unsolicited AEs from the day of vaccination in study V98_06E1 to Day 31. An unsolicited adverse event is an adverse event that was not solicited using a Subject Diary and that was spontaneously communicated by a subject who has signed the informed consent. Potential unsolicited AEs may be medically attended (defined as symptoms or illnesses requiring hospitalization, or emergency room visit, or visit to/by a health care provider), or were of concern to the subject. Possibly Related AE definition: the administration of the investigational vaccine and AE are considered reasonably related in time and the AE could be explained by exposure to the investigational vaccine or by other causes. Probably Related AE definition: exposure to the investigational vaccine and AE are reasonably related in time and no alternative explanation has been identified.
Time Frame: Day 1 to Day 31
Population: All screened subjects who signed informed consent form, provided demographic data and/or baseline screening assessments, were randomized and assigned a study subject ID, received the study vaccination and with any unsolicited adverse event data.
Measure: Count of Participants; unit: Participants
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 14 | 14 | 15 | 10 | 6 | 21
Participants
  Any AE | 4 | 5 | 4 | 4 | 4 | 9
  At least possibly or probably related AEs | 1 | 1 | 0 | 0 | 1 | 1

6. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs), Medically Attended AEs, and AEs Leading to Study Withdrawal
Description: An SAE is defined as any untoward medical occurrence that at any dose results in one or more of the following: Death; life-threatening; that does not refer to an event which hypothetically might have caused death if it were more severe; required or prolonged hospitalization; persistent or significant disability/incapacity; congenital anomaly/or birth defect; any important and significant medical event that may not be immediately life-threatening or resulting in death or hospitalization but, based upon appropriate medical judgement, may jeopardize the subject or may require intervention to prevent one of the other outcomes listed above. "Medically attended adverse event" is defined as an adverse event that leads to a visit to a healthcare provider and "AEs leading to withdrawal" are defined as adverse events leading to study or vaccine withdrawal.
Time Frame: Day 1 to Day 181
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 14 | 14 | 15 | 10 | 6 | 21
Participants
  SAEs | 0 | 0 | 0 | 0 | 0 | 0
  Medically attended AEs | 5 | 5 | 7 | 0 | 2 | 5
  AEs leading to withdrawal | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Subjects With ELISA Antibody Concentrations of GBS Serotype Ia Above Pre-specified Thresholds - Day 31
Description: Percentage of subjects who reach pre-defined sequential serotype-specific serum antibody levels for serotype Ia at Day 31 post-vaccination, as measured by ELISA.
Time Frame: At Day 31
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 13 | 14 | 15 | 10 | 6 | 20
Percentage of subjects
  ≥ 0.1 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [54.1 to 100] | 100 [83.2 to 100]
  ≥ 0.2 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [54.1 to 100] | 85 [62.1 to 96.8]
  ≥ 0.5 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [54.1 to 100] | 80 [56.3 to 94.3]
  ≥ 1 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 83 [35.9 to 99.58] | 75 [50.9 to 91.3]
  ≥ 2 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 67 [22.3 to 95.7] | 60 [36.1 to 80.9]
  ≥ 3 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 67 [22.3 to 95.7] | 60 [36.1 to 80.9]
  ≥ 5 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 93 [68.1 to 99.83] | 90 [55.5 to 99.75] | 67 [22.3 to 95.7] | 60 [36.1 to 80.9]
  ≥ 8 µg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 93 [68.1 to 99.83] | 90 [55.5 to 99.75] | 67 [22.3 to 95.7] | 60 [36.1 to 80.9]

8. Secondary Outcome: Percentage of Subjects With Antibody Concentrations of GBS Serotype Ib Above Pre-specified Thresholds - Day 31
Description: Percentage of subjects who reach pre-defined sequential serotype-specific serum antibody levels for serotype Ib at day 31 post-vaccination. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 31
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 13 | 14 | 15 | 10 | 6 | 20
Percentage of subjects
  ≥ 0.1 μg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [54.1 to 100] | 75 [50.9 to 91.3]
  ≥ 0.2 μg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [54.1 to 100] | 70 [45.7 to 88.1]
  ≥ 0.5 μg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 83 [35.9 to 99.58] | 60 [36.1 to 80.9]
  ≥ 1 μg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 83 [35.9 to 99.58] | 45 [23.1 to 68.5]
  ≥ 2 μg/mL | 100 [75.3 to 100] | 100 [76.8 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 50 [11.8 to 88.2] | 45 [23.1 to 68.5]
  ≥ 3 μg/mL | 100 [75.3 to 100] | 93 [66.1 to 99.82] | 100 [78.2 to 100] | 100 [69.2 to 100] | 50 [11.8 to 88.2] | 45 [23.1 to 68.5]
  ≥ 5 μg/mL | 92 [64 to 99.81] | 93 [66.1 to 99.82] | 100 [78.2 to 100] | 100 [69.2 to 100] | 50 [11.8 to 88.2] | 45 [23.1 to 68.5]
  ≥ 8 μg/mL | 85 [54.6 to 98.1] | 93 [66.1 to 99.82] | 93 [68.1 to 99.83] | 100 [69.2 to 100] | 50 [11.8 to 88.2] | 45 [23.1 to 68.5]

9. Secondary Outcome: Percentage of Subjects With Antibody Concentrations of GBS Serotype III Above Pre-specified Thresholds - Day 31
Description: Percentage of subjects who reach pre-defined sequential serotype-specific serum antibody levels for serotype III at day 31 post-vaccination. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 31
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 13 | 13 | 15 | 10 | 6 | 20
Percentage of subjects
  ≥ 0.1 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 100 [54.1 to 100] | 100 [83.2 to 100]
  ≥ 0.2 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 67 [22.3 to 95.7] | 75 [50.9 to 91.3]
  ≥ 0.5 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 67 [22.3 to 95.7] | 70 [45.7 to 88.1]
  ≥ 1 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 50 [11.8 to 88.2] | 65 [40.8 to 84.6]
  ≥ 2 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 50 [11.8 to 88.2] | 60 [36.1 to 80.9]
  ≥ 3 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 33 [4.3 to 77.7] | 55 [31.5 to 76.9]
  ≥ 5 μg/mL | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [78.2 to 100] | 100 [69.2 to 100] | 33 [4.3 to 77.7] | 55 [31.5 to 76.9]
  ≥ 8 μg/mL | 100 [75.3 to 100] | 92 [64 to 99.81] | 100 [78.2 to 100] | 100 [69.2 to 100] | 33 [4.3 to 77.7] | 50 [27.2 to 72.8]

10. Secondary Outcome: Geometric Mean ELISA Antibody Concentrations of GBS Serotype Ia
Description: The Geometric Mean ELISA Antibody Concentrations of GBS Serotype Ia in All Subjects were estimated for at Day 1, Day 31 and Day 61.
Time Frame: At Day 1, Day 31 and Day 61.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 14 | 14 | 15 | 10 | 6 | 20
µg/mL
  Serotype Ia - Day 1 (V98_06E1) | 9.32 [3.03 to 29] | 5.50 [1.79 to 17] | 3.44 [1.16 to 10] | 2.18 [0.58 to 8.24] | 1.05 [0.19 to 5.86] | 0.32 [0.13 to 0.83]
  Serotype Ia - Day 31: number analyzed (Participants) | 13 | 14 | 15 | 10 | 6 | 20
  Serotype Ia - Day 31 | 61.13 [23 to 165] | 81.61 [31 to 213] | 64.19 [25 to 162] | 57.54 [19 to 179] | 19.25 [4.46 to 83] | 10.06 [4.52 to 22]
  Serotype Ia - Day 61: number analyzed (Participants) | 13 | 14 | 15 | 10 | 5 | 20
  Serotype Ia - Day 61 | 51.53 [21 to 129] | 65.30 [27 to 158] | 44.69 [19 to 105] | 50.67 [18 to 145] | 21.36 [4.85 to 94] | 10.02 [4.77 to 21]

11. Secondary Outcome: Geometric Mean Antibody Concentrations of GBS Serotype Ib
Description: The Geometric Mean Antibody Concentrations of GBS Serotype Ib in All Subjects were estimated for at Day 1, Day 31 and Day 61. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 1, Day 31 and Day 61
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 14 | 14 | 15 | 10 | 6 | 20
µg/mL
  Day 1: number analyzed (Participants) | 14 | 14 | 15 | 10 | 4 | 20
  Day 1 | 0.19 [0.093 to 0.41] | 0.15 [0.073 to 0.32] | 0.10 [0.049 to 0.20] | 0.16 [0.068 to 0.39] | 0.14 [0.035 to 0.55] | 0.17 [0.093 to 0.32]
  Day 31: number analyzed (Participants) | 13 | 14 | 15 | 10 | 6 | 20
  Day 31 | 80.62 [28 to 232] | 74.96 [27 to 207] | 89.59 [33 to 241] | 85.90 [26 to 286] | 6.61 [0.99 to 44] | 3.55 [1.52 to 8.34]
  Day 61: number analyzed (Participants) | 13 | 14 | 15 | 10 | 5 | 20
  Day 61 | 56.32 [22 to 145] | 57.82 [23 to 143] | 59.13 [24 to 143] | 65.53 [22 to 192] | 5.51 [1.01 to 30] | 4.47 [2.09 to 9.58]

12. Secondary Outcome: Geometric Mean Antibody Concentrations of GBS Serotype III
Description: The Geometric Mean Antibody Concentrations of GBS Serotype III in All Subjects were estimated for at Day 1, Day 31 and Day 61. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 1, Day 31 and Day 61
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 14 | 13 | 15 | 10 | 6 | 20
µg/mL
  Day 1: number analyzed (Participants) | 14 | 13 | 15 | 10 | 4 | 20
  Day 1 | 0.41 [0.20 to 0.82] | 0.17 [0.085 to 0.36] | 0.25 [0.13 to 0.49] | 0.17 [0.076 to 0.39] | 0.15 [0.040 to 0.54] | 0.31 [0.17 to 0.55]
  Day 31: number analyzed (Participants) | 13 | 13 | 15 | 10 | 6 | 20
  Day 31 | 111.30 [42 to 294] | 104.55 [40 to 277] | 109.23 [44 to 269] | 216.39 [71 to 655] | 2.66 [0.46 to 15] | 5.33 [2.43 to 12]
  Day 61: number analyzed (Participants) | 13 | 13 | 15 | 10 | 5 | 20
  Day 61 | 91.30 [39 to 214] | 80.94 [34 to 190] | 81.71 [37 to 180] | 200.78 [76 to 531] | 2.67 [0.57 to 12] | 5.82 [2.92 to 12]

13. Secondary Outcome: Geometric Mean ELISA Antibody Concentrations of GBS Serotype Ia in Subjects With Prevaccination Serotype-specific GBS Antibody Less Than the Lower Limit of Quantitation (LLQ)
Description: The Geometric Mean ELISA Antibody Concentrations of GBS Serotype Ia in subjects with prevaccination serotype-specific GBS antibody less than LLQ were estimated for at Day 1, Day 31 and Day 61.
Time Frame: At Day 1, Day 31 and Day 61
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 7 | 10 | 9 | 7 | 4 | 15
µg/mL
  Serotype Ia - Day 1 (V98_06E1) | 1.36 [0.43 to 4.27] | 2.59 [0.99 to 6.75] | 0.81 [0.30 to 2.24] | 1.12 [0.36 to 3.52] | 0.45 [0.099 to 2.05] | 0.16 [0.074 to 0.36]
  Serotype Ia - Day 31 | 32.25 [8.59 to 121] | 62.54 [21 to 189] | 35.47 [11 to 114] | 46.11 [12 to 173] | 6.34 [1.10 to 36] | 3.98 [1.61 to 9.84]
  Serotype Ia - Day 61: number analyzed (Participants) | 7 | 10 | 9 | 7 | 3 | 15
  Serotype Ia - Day 61 | 26.33 [8.12 to 85] | 49.01 [18 to 131] | 24.89 [8.82 to 70] | 39.56 [12 to 128] | 5.79 [0.96 to 35] | 4.25 [1.90 to 9.48]

14. Secondary Outcome: Geometric Mean Antibody Concentrations of GBS Serotype Ib in Subjects With Prevaccination Serotype-specific GBS Antibody Less Than LLQ
Description: The Geometric Mean Antibody Concentrations of GBS Serotype Ib in subjects with prevaccination serotype-specific GBS antibody less than LLQ were estimated for at Day 1, Day 31 and Day 61. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 1, Day 31 and Day 61
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 10 | 9 | 14 | 8 | 3 | 15
µg/mL
  Day 1 | 0.078 [0.078 to 0.078] | 0.078 [0.078 to 0.078] | 0.078 [0.078 to 0.078] | 0.078 [0.078 to 0.078] | 0.078 [0.078 to 0.078] | 0.078 [0.078 to 0.078]
  Day 31 | 60.78 [20 to 182] | 69.05 [22 to 220] | 53.01 [21 to 134] | 65.50 [19 to 224] | 1.47 [0.20 to 11] | 0.79 [0.32 to 1.95]
  Day 61 | 40.59 [15 to 111] | 47.71 [16 to 138] | 34.12 [15 to 80] | 47.58 [15 to 147] | 1.32 [0.21 to 8.37] | 1.19 [0.52 to 2.71]

15. Secondary Outcome: Geometric Mean Antibody Concentrations of GBS Serotype III in Subjects With Prevaccination Serotype-specific GBS Antibody Less Than LLQ
Description: The Geometric Mean Antibody Concentrations of GBS Serotype III in subjects with prevaccination serotype-specific GBS antibody less than LLQ were estimated for at Day 1, Day 31 and Day 61. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 1, Day 31 and Day 61
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 10 | 12 | 11 | 9 | 4 | 15
µg/mL
  Day 1 | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.15] | 0.15 [0.15 to 0.15]
  Day 31 | 109.31 [40 to 301] | 77.97 [31 to 197] | 126.89 [48 to 333] | 188.63 [65 to 549] | 1.90 [0.38 to 9.44] | 2.12 [0.93 to 4.84]
  Day 61 | 83.19 [33 to 208] | 60.01 [26 to 138] | 87.40 [37 to 209] | 169.45 [65 to 444] | 1.92 [0.45 to 8.16] | 2.52 [1.20 to 5.32]

16. Secondary Outcome: Geometric Mean ELISA Antibody Concentrations of GBS Serotype Ia in Subjects With Prevaccination Serotype-specific GBS Antibody Equal or Greater Than LLQ
Description: The Geometric Mean ELISA Antibody Concentrations of GBS Serotype Ia in subjects with prevaccination serotype-specific GBS antibody equal or greater than LLQ were estimated for at Day 1, Day 31 and Day 61.
Time Frame: At Day 1, Day 31 and Day 61
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 7 | 3 | 6 | 2 | 2 | 5
µg/mL
  Serotype Ia - Day 1 (V98_06E1) | 64.06 [23 to 178] | 98.43 [21 to 469] | 29.83 [9.89 to 90] | 39.57 [5.84 to 268] | 5.76 [0.85 to 39] | 2.54 [0.76 to 8.50]
  Serotype Ia - Day 31: number analyzed (Participants) | 6 | 3 | 6 | 2 | 2 | 5
  Serotype Ia - Day 31 | 128.91 [71 to 234] | 196.32 [85 to 456] | 156.26 [86 to 284] | 85.63 [31 to 240] | 177.38 [63 to 498] | 161.99 [84 to 311]
  Serotype Ia - Day 61: number analyzed (Participants) | 6 | 3 | 6 | 2 | 2 | 5
  Serotype Ia - Day 61 | 112.78 [57 to 222] | 197.67 [76 to 515] | 107.57 [55 to 212] | 93.02 [29 to 300] | 151.27 [47 to 488] | 131.48 [63 to 276]

17. Secondary Outcome: Geometric Mean Antibody Concentrations of GBS Serotype Ib in Subjects With Prevaccination Serotype-specific GBS Antibody Equal or Greater Than LLQ
Description: The Geometric Mean Antibody Concentrations of GBS Serotype Ib in subjects with prevaccination serotype-specific GBS antibody equal or greater than LLQ were estimated for at Day 1, Day 31 and Day 61. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 1, Day 31 and Day 61
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 4 | 5 | 1 | 2 | 1 | 5
µg/mL
  Day 1 | 1.96 [0.56 to 6.85] | 0.52 [0.17 to 1.60] | 3.42 [0.28 to 42] | 3.12 [0.53 to 18] | 0.82 [0.067 to 10] | 1.92 [0.63 to 5.89]
  Day 31: number analyzed (Participants) | 3 | 5 | 1 | 2 | 1 | 5
  Day 31 | 287.34 [90 to 917] | 121.26 [44 to 333] | 373.02 [48 to 2877] | 338.80 [78 to 1469] | 557.46 [75 to 4142] | 557.03 [225 to 1379]
  Day 61 | 228.26 [72 to 726] | 118.94 [43 to 326] | 367.26 [48 to 2818] | 300.10 [69 to 1296] | 378.70 [51 to 2800] | 403.16 [163 to 996]

18. Secondary Outcome: Geometric Mean Antibody Concentrations of GBS Serotype III in Subjects With Prevaccination Serotype-specific GBS Antibody Equal or Greater Than LLQ
Description: The Geometric Mean Antibody Concentrations of GBS Serotype III in subjects with prevaccination serotype-specific GBS antibody equal or greater than LLQ were estimated for at Day 1, Day 31 and Day 61. As the singleton ELISA was no longer in use at the time of serotypes Ib and III testing, results for both serotypes were tested using multiplex immunoassay.
Time Frame: At Day 1, Day 31 and Day 61
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 4 | 1 | 4 | 1 | 0 | 5
µg/mL
  Day 1 | 5.33 [0.76 to 37] | 1.41 [0.029 to 68] | 1.07 [0.15 to 7.46] | 0.74 [0.015 to 36] |  | 2.79 [0.49 to 16]
  Day 31: number analyzed (Participants) | 3 | 1 | 4 | 1 | 0 | 5
  Day 31 | 171.67 [13 to 2214] | 270.01 [3.46 to 21064] | 120.00 [13 to 1113] | 149.93 [1.81 to 12454] |  | 136.68 [19 to 979]
  Day 61: number analyzed (Participants) | 3 | 1 | 4 | 1 | 0 | 5
  Day 61 | 186.63 [24 to 1439] | 231.17 [7.12 to 7509] | 107.21 [18 to 635] | 180.29 [5.28 to 6158] |  | 116.43 [24 to 561]

19. Secondary Outcome: Geometric Mean ELISA Anti-Diphtheria Antibody Concentrations in All Subjects
Description: Geometric Mean ELISA Anti-Diphtheria Antibody Concentrations (95%CI) in All Subjects at Day 1 Pre-vaccination in the V98_06 study or V98_06E1 for the Naive Group and at Day 61 Post-vaccination in Study V98_06E1. Anti-diphtheria antibody testing was not performed in this study because no diphtheria vaccine was administered in the study and also because data from other Cross Reactive Material(CRM)-based vaccines demonstrate that administration has not resulted in a decline in anti-diphtheria antibody concentrations.
Time Frame: At Day 1 (V98_06 or V98_06E1) and Day 61
Population: Anti-diphtheria antibody testing was not performed in this study because no diphtheria vaccine was administered in the study and also because data from other CRM-based vaccines demonstrate that administration has not resulted in a decline in anti-diphtheria antibody concentrations.
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected until 7 days after vaccination. Unsolicited AEs were collected from Day 1 to Day 181. SAEs were collected from Day 1 to Day 181.
Arm/Group | GBS NoAdj/GBS NoAdj Group | GBS Alum/GBS NoAdj Group | GBS MF59 Half/GBS NoAdj Group | GBS MF59 Full/GBS NoAdj Group | Placebo/GBS NoAdj Group | Naive/GBS NoAdj Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/15 | 0/10 | 0/6 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/15 | 0/10 | 0/6 | 0/21
Other Adverse Events (participants affected / at risk) | 13/14 | 13/14 | 13/15 | 7/10 | 4/6 | 17/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GBS NoAdj/GBS NoAdj Group (N=14) | GBS Alum/GBS NoAdj Group (N=14) | GBS MF59 Half/GBS NoAdj Group (N=15) | GBS MF59 Full/GBS NoAdj Group (N=10) | Placebo/GBS NoAdj Group (N=6) | Naive/GBS NoAdj Group (N=21)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (11) | 10 (13) | 4 (9) | 4 (6) | 1 (3) | 2 (2)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (3) | 4 (6) | 2 (2) | 1 (1) | 1 (8) | 3 (5)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Injection site induration (General disorders) | 2 (3) | 2 (3) | 5 (10) | 2 (6) | 1 (5) | 0 (0)
Injection site pain (General disorders) | 10 (20) | 9 (15) | 9 (19) | 6 (10) | 3 (12) | 11 (23)
Injection site swelling (General disorders) | 0 (0) | 2 (3) | 4 (6) | 1 (3) | 1 (5) | 0 (0)
Injection site warmth (General disorders) | 1 (2) | 4 (5) | 4 (7) | 2 (3) | 2 (8) | 2 (2)
Malaise (General disorders) | 0 (0) | 2 (3) | 2 (3) | 2 (3) | 1 (1) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (3) | 3 (4) | 1 (1) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (12) | 6 (12) | 5 (9) | 3 (3) | 2 (4) | 4 (6)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hangover (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT02690181/Prot_SAP_000.pdf